CLINICAL TRIAL: NCT03543514
Title: STUDY ON THE EFFECT OF TRIMODAL PREHABILITATION IN PATIENTS SUBMITTED TO RECTAL SURGERY DURING ADJUVANCY OR BEFORE SURGERY
Brief Title: PREHABILITATION RECTAL CANCER DURING ADJUVANCY VS BEFORE SURGERY
Acronym: prehab-cspt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Laura Mora-Lopez, DOCTOR, Corporacion Parc Tauli
Other Study IDs: PREHAB-CSPT
Record Dates: First submitted 2018-04-26; First posted 2018-06-01 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Colo-rectal Cancer
Keywords: colon cancer, rectal cancer, prehabilitation
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PREHABILITATION GROUP: Patients affected on Cold-rectal cancer who needs surgery. We made trimodal prehabilitation
  Interventions: Other: TRIMODAL PREHABILITATION

INTERVENTIONS:
Other: TRIMODAL PREHABILITATION — Trimodal prehabilitation application in the form of:
  * Control with the 6-minute walking test and podometer of physical activity
  * Dietary advice to be able to perform a hyperproteic diet
  * Mindfullnes to improve the emotional level.
  Other Names: PHYSICAL INTERVENTION; NUTRITIONAL INTERVENTION; EMOTIONAL INTERVENTION

SUMMARY:
Preoperative preparation protocol (prehabilitation) for patients diagnosed with colorectal cancer who need surgery. It consists of a change in the preoperative preparation. The patient is an active part of their preparation and the professionals help to achieve a better functional capacity to diminish morbidity and accelerate recovery. Three levels are controlled:

* Physical: control and stimulation to exercise at home.
* Nutrition: control and advice through homemade recipes.
* Emotional: control of the level of haste or depression and advice of mindfullness techniques at home.

If they need specific help they are derived from specialized professionals (rehabilitator, nutritionist / endocrinologist, psychologist).

DETAILED DESCRIPTION:
Protocol for colorectal neoplasia patients who need surgery by modifying the current one. Until now, in the preoperative time, the anesthetist evaluated the need for some specific action such as pre-operative iron administration to avoid perioperative transfusions or the need to assess some of the patient's morbidities to try to optimize it. In the perioperative period in our hospital, the criteria of the Multimodal and Fast-Tcack Rehabilitation programs have been applied for a long time and there are some trajectories that allow standardization of patient management once they have been admitted.

It is demonstrated in other centers and in other surgical pathologies that, in addition to what we are already applying to our center, modify the preoperative preparation of our patients and try to improve their "functional capacity" results of lower morbidity and mortality and the subsequent recovery of patients can greatly improve . This is called prehabilitation. Pretreatment consists in a change in preoperative preparation at three levels. The concept of preoperative preparation changes and the patient is actively involved in it. Three levels of the patient are controlled: functional or physical level, nutritional level and emotional level, by means of pots and they are encouraged to make a series of changes in their habitual life (exercise, dietary advice, mindfullness techniques) that increase its functional capacity. This is related to a decrease in morbidity and mortality and in addition to a better and faster postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with colorectal neoplasia
* Need colorectal surgery with curative indication
* Scheduled surgery

Exclusion Criteria:

* Patients who refuse to enter the study
* Patients with indication of palliative surgery
* Surgeries that involve colon and other organs
* Urgent surgery
* Basic pathology that does not allow to carry out some of the explorations necessary to carry out the trimodal pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by a colon or rectal tumor that have to undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Crompehension Complexity Index (CCI) | 30 days
  General morbidity due to the improvement of the physical capacity, the nutritional profile and the diminution of the psychic stroke can be diminished throughout the process and the return to the basal situation.

SECONDARY OUTCOMES:
Six minutes walking test (6-MWT) | 30 days
  Physical capacity
Malnutrion Universal Screening Tool (MUST) | 30 days
  Nutritional condition
Hospital Anxiety and Depression Scale (HADS) | 30 days
  Emotional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mora, Dr., Principal Investigator — Hospital Universitari Parc Tauli
Locations (2):
- Spain (2):
  - Laura Mora López, Sabadell, Barcelona
  - Laura Mora Löpez, Sabadell, Barcelona

IPD SHARING:
Plan to Share IPD: No
There's no plan to share IPD to other researchers

REFERENCES:
- [Background] Zingmond D, Maggard M, O'Connell J, Liu J, Etzioni D, Ko C. What predicts serious complications in colorectal cancer resection? Am Surg. 2003 Nov;69(11):969-74. PMID 14627258
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Christensen T, Kehlet H. Postoperative fatigue. World J Surg. 1993 Mar-Apr;17(2):220-5. doi: 10.1007/BF01658930. PMID 8511917
- [Background] Carli F, Mayo N, Klubien K, Schricker T, Trudel J, Belliveau P. Epidural analgesia enhances functional exercise capacity and health-related quality of life after colonic surgery: results of a randomized trial. Anesthesiology. 2002 Sep;97(3):540-9. doi: 10.1097/00000542-200209000-00005. PMID 12218518
- [Background] Carli F, Zavorsky GS. Optimizing functional exercise capacity in the elderly surgical population. Curr Opin Clin Nutr Metab Care. 2005 Jan;8(1):23-32. doi: 10.1097/00075197-200501000-00005. PMID 15585997
- [Background] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Background] Lawrence VA, Hazuda HP, Cornell JE, Pederson T, Bradshaw PT, Mulrow CD, Page CP. Functional independence after major abdominal surgery in the elderly. J Am Coll Surg. 2004 Nov;199(5):762-72. doi: 10.1016/j.jamcollsurg.2004.05.280. PMID 15501119
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Background] Burden ST, Hill J, Shaffer JL, Todd C. Nutritional status of preoperative colorectal cancer patients. J Hum Nutr Diet. 2010 Aug;23(4):402-7. doi: 10.1111/j.1365-277X.2010.01070.x. Epub 2010 May 13. PMID 20487172
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Leon-Pizarro C, Gich I, Barthe E, Rovirosa A, Farrus B, Casas F, Verger E, Biete A, Craven-Bartle J, Sierra J, Arcusa A. A randomized trial of the effect of training in relaxation and guided imagery techniques in improving psychological and quality-of-life indices for gynecologic and breast brachytherapy patients. Psychooncology. 2007 Nov;16(11):971-9. doi: 10.1002/pon.1171. PMID 17311247
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682